CLINICAL TRIAL: NCT06423378
Title: Bio-Integrative, Fiber-Reinforced Kneebar for Treating Subchondral Insufficiency of the Knee
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Lance LeClere, Dr. Lance LeClere, MD; Principal Investigator, Associate Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSSIOfiber Kneebar
Record Dates: First submitted 2024-05-07; First posted 2024-05-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Subchondral Insufficiency Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: OSSIOfiber® Trimmable Fixation Nails — Subjects will be treated with cannulated nails before or after arthroscopic management of their concomitant pathology at the discretion of the investigator. Technique described below. Following nail placement, tissue layers will be closed in standard fashion.
  1. Preop MRI views used to estimate the proper depth & location of nail placement on the femur and/or tibia
  2. Exposure is gained to medial tibia
  3. 1.4 mm K-Wire is placed through medial tibia parallel to the articular joint surface ~ 1 cm distal to the articular joint line
  4. A depth gauge is placed over K-Wire to determine required length of cannulated nail
  5. A 4.0 mm cannulated drill bit used over K-Wire to prepare the pilot hole
  6. Tamp is used to insert pre-trimmed 4.0 mm cannulated nail into the pilot hole and K-Wire is subsequently removed
  7. Intraop fluoroscopy can confirm adequate nail placement prior to removing K-wire
  8. Repeat steps for additional nails

SUMMARY:
The OSSIOfiber® Trimmable Fixation Nails are indicated for maintenance of alignment and fixation of bone fractures, osteotomies, arthrodesis and bone grafts in the presence of appropriate additional immobilization (e.g., rigid fixation implants, cast, brace). Our hypothesis is that the use of OSSIOfiber® Trimmable Fixation Nails for treating subchondral insufficiency of the knee will result in improvement of patient-reported outcomes and imaging findings. The primary objective of this study is to evaluate the effectiveness of implanting bio-integrative OSSIOfiber® Trimmable Fixation Nails, organized in a bi-cortical rafter formation within the tibia or femur for the management of subchondral insufficiency. The OSSIOfiber® Trimmable Fixation Nails used in this study will be considered on-label.

ELIGIBILITY:
Inclusion Criteria:

* Agree to study participation and consent obtained.
* Able to attend all postoperative clinical visits, undergo imaging procedures, and complete relevant questionnaires.
* Subjects between the ages of 18 to 75 years.
* Body Mass Index < 40.
* Has knee pain in the study knee lasting at least 3 months and has had at least moderate pain recorded on a standard of care (SOC) preoperative Knee Injury and Osteoarthritis Outcome Score (KOOS) and/or Numeric Pain Reported Scale (0-10) questionnaire. The study team may utilize these verbal pain scores collected during the clinic intake process for screening purposes. If the patient was not administered the verbal pain score, the patient will be consented, administered the pain survey, and withdrawn if moderate pain score was not recorded.
* At least 3-months without steroid injection or any other non-surgical intervention administered to study knee.
* Candidate for knee arthroscopy due to meniscal tear, loose body, unstable articular cartilage or mechanical symptoms.
* Uni-compartmental Kellgren-Lawrence grade 2-3 osteoarthritis in the study tibia or femur.
* Bone Marrow Lesion (BML) confirmed on magnetic resonance imaging in the femur, tibia or both.
* Cartilage lesion on the tibial or femoral condyle(s) of a grading ≤4 by either the International Cartilage Repair Society or Outerbridge classifications verified at the time of arthroscopy.

Exclusion Criteria:

* Imaging evidence of the study knee that includes any of the following:

  1. Kellgren-Lawrence grade 4 osteoarthritis.
  2. Collapse of subchondral bone.
  3. Avascular Necrosis (AVN).
  4. Osteochondral defect overlying the BML
  5. BML located at ACL or PCL insertions
* Clinical evidence of the study knee that includes any of the following:

  1. History of rheumatoid arthritis, septic arthritis, reactive arthritis, gout or pseudogout, secondary arthropathy (e.g., hemochromatosis, hemophilia, or psoriasis).
  2. Osteochondritis dissecans.
  3. Frank ligamentous instability.
  4. Neuromuscular deficiency or other that would limit the ability to do a functional assessment.
* Bi-cortical nail implantation cannot be achieved, including where the required nail length is not yet available.
* Current tobacco use or has quit within 3 months of study enrolment.
* Substance abuse history.
* Diabetes mellitus, HbA1c>8
* High surgical risk due to pre-existing conditions.
* Currently pregnant or has plans to become pregnant prior to surgery.
* Active infection or history of chronic infection in study knee.
* Will require concomitant procedures within study knee, including but not limited to ligament reconstruction, tendon repair, meniscus repair, microfracture, osteotomy, or osteochondral transplantation (Meniscal tears, including chronic, are acceptable if no repair is required)
* Significant malalignment (varus or valgus) of the knee (>8°)
* Use of augmentation or concomitant biologic therapy during surgery.
* Contraindications to magnetic resonance imaging.
* Any condition which in the view of the treating physician makes it inadvisable for the subject to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 3 months post-operatively
  The overall KOOS score combines pain and function domains. KOOS is out 100, where 0 equates to extreme pain and 100 equates to no pain.
Knee injury and Osteoarthritis Outcome Scale Score (KOOS) | 6 months post-operatively
  The overall KOOS score combines pain and function domains. KOOS is out 100, where 0 equates to extreme pain and 100 equates to no pain.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | 6 months post-operatively
  Measures the knee health of individuals following surgery
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form | 6 months post-operatively
  IKDC measures: symptoms, athletic activity, and knee function.
Veterans Rand-12 (VR-12) Health Survey Scale Score | 6 months post-operatively
  VR-12 combines measures of general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, fatigue , social functioning, and mental health
Numeric Pain Reported Scale Score | 6 months post-operatively
  Measures a subject's perceived pain level. This score is usually on a scale of 0-10 with 0 equating to no pain and 10 equating to the worst pain imaginable.
PROMIS Pain Interference Score | 6 months post-operatively
  Measures what level pain hinders a patient's engagement in several activities including social, cognitive, physical, and recreational activities. There are 7 sub items and each are rated from a scale of 0-10 where 0 means it does not interfere and 10 means it completely interferes. These contribute to a final score ranging anywhere from 0-70.
PROMIS Depression Score | 6 months post-operatively
  Measures self-reported negative mood (sadness, guilt), views of self (self- criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40. Higher scores indicate greater severity of depression.
PROMIS Physical Function Score | 6 months post-operatively
  Measures the level of physical function for patients with a wide variety of impairments that may limit the patient's physical capability. This score is on a scale from 0-100 with 0 equating to no physical function and 100 equating to optimal physical function.
Incidence Assessments | Up to 6 month post-operatively
  Assessment of the incidence of re-operations, revision surgeries, or additional management of the study knee outside of postoperative rehabilitation.
Degree of knee ligament healing | Baseline and 6 months post-operatively
  To see how the knee ligament is healing by MRI assessment.
Adverse Events | Up to 6 month post-operatively
  Rate of postoperative adverse events and complications

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No